CLINICAL TRIAL: NCT02614846
Title: A Safety, Pharmacokinetics and Pharmacodynamics Study of Hetrombopag Olamine in Chronic Idiopathic Thrombocytopenic Purpura
Brief Title: Safety and Efficacy Study of Hetrombopag Olamine in Chronic Idiopathic Thrombocytopenic Purpura (ITP) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-TPO- Ie-ITP
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura

ARMS (1):
- Hetrombopag Olamine (Experimental): All the subjects receive 6 weeks Hetrombopag Olamine dosing, 5mg for the first 2 weeks, 2.5mg or 7.5mg for the last 4 weeks according to the PLT counting.
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine

SUMMARY:
This study evaluates the safety and efficacy of 6 weeks dosing Hetrombopag Olamine in Chronic Idiopathic Thrombocytopenic Purpura Patients. All of the subjects in this study receive Hetrombopag.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Confirmed diagnosis of chronic ITP,a peripheral blood smear or bone marrow examination should support the diagnosis of ITP with no evidence of other causes of thrombocytopenia.
  2. Patients had a platelet count of less than 30,000/µL both in the screening period and baseline.
  3. Subjects who are refractory or have relapsed after at least one prior ITP therapy.
  4. Previous therapy for ITP including rescue must have been completed at least 2 weeks prior to randomization.
  5. Subjects treated with maintenance immunosuppressive therapy must be receiving a dose that has been stable for at least 1 month.
  6. A complete blood count (CBC), within the reference range, with the following exceptions.
* Platelets <30×109/L is required for inclusion .
* Hemoglobin: females and males 10.0 g/dl are eligible for inclusion.
* Absolute neutrophil count (ANC) ≥1500/µL (1.5×109/L) is required for inclusion.

  7.PT result no exceed normal by more than ±3s,APTT result no exceed normal by more than ±10s.

  8.Female subjects have a negative result with HCG testing in the screening period and baseline.
* Exclusion Criteria:

  1. Patients with any prior history of arterial or venous thrombosis，or diagnosis as Thrombophilia.
  2. Subjects diagnosed with tumor.
  3. Have pre-existing cardiac disease within the last 3 months.No arrhythmia known to increase the risk of thrombolic events (e.g. atrial fibrillation), or patients with a Corrected QT interval (QTc) >450msec or QTc >480 for patients with a Bundle Branch Block.
  4. Female subjects who are nursing or pregnant at screening or pre-dose on baseline.
  5. Treatment with thrombopoietin or an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
  6. Treatment with Rituximab or Splenectomy within the lat 6 months.
  7. Subjects who have previously received eltrombopag or any other thrombopoietin receptor agonist within 30 days or five half-lives (whichever is longer).
  8. Subject has consumed aspirin, aspirin-containing compounds, salicylates, anticoagulants, quinine or non-steroidal anti-inflammatories (NSAIDs) for >3 consecutive days within 2 weeks of the study start and until the end of the study.
  9. Any laboratory or clinical evidence for HIV infection.Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subject screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with adverse events as a measure of safety and tolerability. | From Day 1 to Day 70.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and technology, Wuhan, Hubei, China